CLINICAL TRIAL: NCT02463864
Title: A Randomised Controlled Trial to Measure the Effects of Twice-Daily Individual, Targeted, Strengthening, Balance and Endurance Exercise Sessions on Mobility, Quality of Life and Healthcare Utilisation for Frail Older Medical In-patients
Brief Title: A Twice-Daily Individual Targeted Exercise Program in Frail Hospitalised Older Medical In-patients (RCT)
Acronym: APEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr Suzanne Timmons, Senior Lecturer in Gerontology and Rehabilitation, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCCork
Record Dates: First submitted 2015-05-26; First posted 2015-06-04 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Frail Older Adults
Keywords: frailty; older adult; hospital; exercise; randomised control trial; functional decline
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention exercise (Experimental): Twice daily, individual, targeted, strengthening, balance and endurance exercise sessions
  Interventions: Other: Intervention exercise
- Sham exercise (Sham Comparator): Twice daily, individual, stretching and relaxation exercise sessions
  Interventions: Other: Sham Exercise

INTERVENTIONS:
Other: Intervention exercise — Twice daily, individual, targeted, strengthening, balance and endurance exercises for the duration of the hospital stay, prescribed and delivered by a senior physiotherapist.
  Other Names: Augmented Prescribed Exercise Program
  Arms: Intervention exercise
Other: Sham Exercise — Twice daily stretching and relaxation exercises for the duration of the hospital stay, by a senior physiotherapist.
  Arms: Sham exercise

SUMMARY:
This study will help to determine whether frail older medical inpatients will benefit from targeted exercise sessions performed twice daily while in hospital. Half of the patients will complete targeted strengthening, balance and endurance exercises and the other half, stretching and relaxation exercises. The exercise sessions will be assisted and supported by a senior physiotherapist.

DETAILED DESCRIPTION:
It is well known that older medical patients can experience functional decline following an acute hospital admission and this can persist for up to three months. The targeted exercises are designed to prevent this functional decline by maintaining the patients' strength, balance and endurance. To counterbalance the considerable time spent with the physiotherapy services in the intervention arm, the control group will receive stretches and relaxation exercises. Patients' length of stay is the primary outcome measure. Their physical performance and quality of life at discharge and at 3 months post discharge and their readmission rates are the secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* medical patients
* anticipated length of stay greater than 2 days
* planned for discharge home
* mobility aid and /or assistance required on admission

Exclusion Criteria:

* contraindications to exercise
* unable to follow commands in the English language
* unable to exercise with the assistance of one person only
* when active palliative care is required
* when full isolation for containment of a contagious infection is required

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Length of Stay | At time of discharge from hospital (an expected average of 8 days post admission)
  Patients length of hospital stay is recorded at the time of discharge from electronic admissions data

SECONDARY OUTCOMES:
Physical Performance | At time of discharge from hospital (an expected average of 8 days post admission); and again at 3 months post discharge
  The Short Physical Performance Battery will be completed, which includes a timed 4 m walk. Patients can score 0-12; scoring higher with better physical performance.
Quality of Life | At time of discharge from hospital (an expected average of 8 days post admission); and again at 3 months post discharge
  The EQ5D-5L will be completed by the patient.
Re-admission Rate | From the time of hospital discharge to 3 months post discharge
  The number of admissions within 3 months following the index admission will be recorded from hospital electronic records

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Timmons, Principal Investigator — University College Cork
Locations (1):
- Mercy University Hospital, Cork, Ireland

REFERENCES:
- [Derived] McCullagh R, O'Connell E, O'Meara S, Dahly D, O'Reilly E, O'Connor K, Horgan NF, Timmons S. Augmented exercise in hospital improves physical performance and reduces negative post hospitalization events: a randomized controlled trial. BMC Geriatr. 2020 Feb 7;20(1):46. doi: 10.1186/s12877-020-1436-0. PMID 32033532
- [Derived] McCullagh R, O'Connell E, O'Meara S, Perry I, Fitzgerald A, O'Connor K, Horgan NF, Timmons S. A study protocol of a randomised controlled trial to measure the effects of an augmented prescribed exercise programme (APEP) for frail older medical patients in the acute setting. BMC Geriatr. 2016 Apr 8;16:79. doi: 10.1186/s12877-016-0252-z. PMID 27059306